CLINICAL TRIAL: NCT04142437
Title: PrOspective Non-interventional Study in Patients With Locally Advanced or Metastatic TRK Fusion Cancer Treated With Larotrectinib
Brief Title: Study to Learn More About the Safety and Effectiveness of the Drug VITRAKVI During Routine Use in Patients With TRK Fusion Cancer Which is Locally Advanced or Spread From the Place Where it Started to Other Places in the Body
Acronym: ON-TRK
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20324
Record Dates: First submitted 2019-10-17; First posted 2019-10-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced or Metastatic Solid Tumor Harboring an NTRK Gene Fusion
MeSH Terms: interventions — larotrectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (8):
- GI: adult patients with gastrointestinal (GI) cancer
  Interventions: Drug: larotrectinib(Vitrakvi, BAY2757556)
- H&N: adult patients with head and neck (H&N) cancer
  Interventions: Drug: larotrectinib(Vitrakvi, BAY2757556)
- STS: adult patients with soft tissue sarcoma (STS)
  Interventions: Drug: larotrectinib(Vitrakvi, BAY2757556)
- CNS: adult patients with primary central nervous system (CNS) cancer
  Interventions: Drug: larotrectinib(Vitrakvi, BAY2757556)
- Lung: adult patients with lung cancer
  Interventions: Drug: larotrectinib(Vitrakvi, BAY2757556)
- Melanoma: adult patients with melanoma
  Interventions: Drug: larotrectinib(Vitrakvi, BAY2757556)
- Pediatric: all pediatric patients regardless of tumor type will be enrolled under this cohort
  Interventions: Drug: larotrectinib(Vitrakvi, BAY2757556)
- other: patients with other tumor types
  Interventions: Drug: larotrectinib(Vitrakvi, BAY2757556)

INTERVENTIONS:
Drug: larotrectinib(Vitrakvi, BAY2757556) — In the study, patients treated under local standard of care clinical practice; all decisions in terms of diagnostic procedures, treatments, management of the disease, and resource utilization are fully dependent on mutual agreement between the patient and the attending physician, without interference by the study initiator or study protocol

SUMMARY:
In this observational study researcher want to learn more about the effectiveness of drug VITRAKVI (generic name: larotrectinib) and how well the drug is tolerated during routine use in patients with TRK fusion cancer which is locally advanced or spread from the place where it started to other places in the body. TRK fusion cancer is a term used to describe a variety of common and rare cancers that are caused by a change to the NTRK (Neurotrophic Tyrosine Kinase) gene called a fusion. During this fusion, an NTRK gene joins together, or fuses, with a different gene. This joining results in the activation of certain proteins (TRK fusion proteins), which can cause cancer cells to multiply and form a tumor. VITRAKVI is an approved drug that blocks the action of the NTRK gene fusion. This study will enroll adult and paediatric patients suffering from a solid tumor with NTRK gene fusion for whom the decision to treat their disease with VITRAKVI has been made by their treating physicians. During the study, patients' medical information such as treatment information with VITRAKVI, other medication or treatments, changes in disease status and other health signs and symptoms will be collected within the normal medical care by the treating doctor. Participants will be observed over a period from 24 to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric (from birth to 18-year-old) patients
* Patients with locally advanced or metastatic solid tumor harboring an NTRK gene fusion. NTRK (NTRK1, NTRK2, and NTRK3) gene fusions will be identified locally. Acceptable methods of detection of NTRK gene fusion include NGS, fluorescence in situ hybridization (FISH), reverse-transcription polymerase chain reaction (rt-PCR) or any other genomic testing able to detect NTRK gene fusion. If a pan-TRK IHC method is used, this result needs to be accompanied with the results using one of the other methods noted above.
* Life expectancy of at least 3 months based on clinical judgement
* Decision to treat with larotrectinib made by the treating physician prior to study enrollment
* Patients can also be enrolled if the initial visit (larotrectinib start date) occurred within 2 months ±3 days prior to informed consent signed date
* Signed informed consent form
* For patients under legal age, signed assent by the patient (where applicable) and parental/legal guardian signed informed consent is required

Exclusion Criteria:

* Any contraindications as listed in the local approved product information
* Pregnancy
* Participation in an investigational program with interventions outside of routine clinical practice
* Prior treatment with larotrectinib or other kinase inhibitor with TRK inhibition
* Patients with NTRK gene amplification or NTRK point mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric (from birth to 18-year-old) patients with a locally advanced or metastatic solid tumor harboring an NTRK gene fusion (detected by NGS (Next-Generation Sequencing), FISH (Fluorescent In Situ Hybridization), rt-PCR (Reverse Transcription Polymerase Chain Reaction) or other genomic testing able to detect NTRK gene fusion) assessed locally for whom a decision to treat with larotrectinib has been made before enrollment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 30 days after last dose
Severity of TEAEs | Up to 30 days after last dose
Seriousness of TEAEs | Up to 30 days after last dose
Reasonable causal relationship between larotrectinib and an AE | Up to 30 days after last dose
Causality of TEAEs | Up to 30 days after last dose
Action taken related to larotrectinib treatment | Up to 30 days after last dose

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 8 years
Disease control rate (DCR) | Up to 8 years
Duration of response (DOR) | Up to 8 years
Time to response (TTR) | Up to 8 years
Progression-free survival (PFS) | Up to 8 years
Overall survival (OS) | Up to 8 years
Total dose | Up to 8 years
Starting and ending dose | Up to 8 years
Dose modification during treatment | Up to 8 years
Duration of treatment (DOT) | Up to 8 years
ORR by patient subgroup(s) | Up to 8 years
DCR by patient subgroup(s) | Up to 8 years
DOR by patient subgroup(s) | Up to 8 years
TTR by patient subgroup(s) | Up to 8 years
PFS by patient subgroup(s) | Up to 8 years
OS by patient subgroup(s) | Up to 8 years
Number of patients with change in height and weight from baseline by visit, neurological abnormalities (normal/abnormal) | Up to 8 years
  for all patients
Number of patients with abnormal developmental milestones | Up to 8 years
  Pediatric cohort only
Number of patients with abnormal Tanner stage | Up to 8 years
  Pediatric cohort only

CONTACTS AND LOCATIONS:
Locations (76):
- United States (51):
  - Banner Desert Medical Center, Mesa, Arizona
  - California Research Inst., Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA - Mattel Children's Hospital, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Stanford Univ Med Ctr. / Lucile Packard Children's Hosp, Palo Alto, California
  - Providence Health System - Southern California, Santa Monica, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - SCL Health, Grand Junction, Colorado
  - Yale University, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Fort Wayne Medical Oncology Hematology, Fort Wayne, Indiana
  - Regional Health Hope Center, Terre Haute, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Maine Health, South Portland, Maine
  - Univ. of Maryland / Greenebaum Comp. Cancer Ctr., Baltimore, Maryland
  - Johns Hopkins / Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Frederick Health-James M Stockman Cancer Institute, Frederick, Maryland
  - Tufts / Neely Cancer Center, Boston, Massachusetts
  - Boston Children's / Dana Farber, Boston, Massachusetts
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Sparrow Cancer Center, Lansing, Michigan
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Atlantic Hem Onc / Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Great Lakes Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Children's Cancer Center, New York, New York
  - Staten Island Univ. Hospital (Northwell Health), Staten Island, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - East Carolina University / Vidant Health, Greenville, North Carolina
  - Ohio State Comp. Cancer Ctr. / James Cancer Hospital, Columbus, Ohio
  - Mercy Health Youngstown, Youngstown, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania (Penn Med), Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Medical Univ. of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center / Children's Health, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Intermountain Healthcare - Intermountain Medical Center, Murray, Utah
  - Univ. of Utah / Huntsman Cancer Center, Salt Lake City, Utah
  - Intermountain Healthcare - Dixie Regional Medical Center, St. George, Utah
  - Seattle Children's, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Gundersen Health System, La Crosse, Wisconsin
  - SSM Health Cancer Center - Dean Medical Group, Madison, Wisconsin
- Many Locations, Multiple Locations, Argentina
- Many Locations, Multiple Locations, Australia
- Many Locations, Multiple Locations, Austria
- Many Locations, Multiple Locations, Belgium
- Many Locations, Multiple Locations, Brazil
- Many Locations, Multiple Locations, Canada
- Many Locations, Multiple Locations, China
- Many Locations, Multiple Locations, Denmark
- Many Locations, Multiple Locations, Finland
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Greece
- Many Locations, Multiple Locations, Ireland
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Japan
- Many Locations, Multiple Locations, Luxembourg
- Many Locations, Multiple Locations, Norway
- Many Locations, Multiple Locations, Russia
- Many Locations, Multiple Locations, Singapore
- Many Locations, Multiple Locations, South Korea
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Sweden
- Many Locations, Multiple Locations, Switzerland
- Many Locations, Multiple Locations, Taiwan
- Many Locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Yang JCH, Brose MS, Castro G, Kim ES, Lassen UN, Leyvraz S, Pappo A, Lopez-Rios F, Reeves JA, Fellous M, Penault-Llorca F, Rudzinski ER, Tabatabai G, Vassal G, Drilon A, Trent J. Rationale and design of ON-TRK: a novel prospective non-interventional study in patients with TRK fusion cancer treated with larotrectinib. BMC Cancer. 2022 Jun 7;22(1):625. doi: 10.1186/s12885-022-09687-x. PMID 35672677
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/